CLINICAL TRIAL: NCT02173041
Title: Impact of Prevention Awareness Group (PAG) on Treatment Attendance and Drug Abstinence Among Substance User: Results of the Randomized Controlled Trial
Brief Title: Impact of Prevention Awareness Group (PAG) on Treatment Attendance and Drug Abstinence Among Substance User
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Macmillan Research Group UK (Industry)
Collaborators: NMP Medical Research Institute (Other); Warwick Research Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mac/NMP 1216
Record Dates: First submitted 2014-06-22; First posted 2014-06-24 (Estimated); Last update posted 2015-05-18 (Estimated); Status verified 2015-05

CONDITIONS: Substance Use Disorder; Drug Dependence,; Alcohol Dependence
Keywords: Prevention and Awareness Groups (PAG),; Substance Use Disorder,; Community based intervention
MeSH Terms: conditions — Substance-Related Disorders; Alcoholism | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Usual Care (Other): Community program which follows with referral services
  Interventions: Other: Standard Care
- Prevention Awareness Groups (PAG) (Experimental): Prevention Awareness Groups (PAG) is a community based integrated substance abuse prevention program targeting vulnerable populations. It comprises of community programs, physician led counseling followed by treatment follow up in community based clinic.
  Interventions: Other: Prevention Awareness Groups (PAG)

INTERVENTIONS:
Other: Prevention Awareness Groups (PAG)
  Arms: Prevention Awareness Groups (PAG)
Other: Standard Care
  Arms: Standard Usual Care

SUMMARY:
Substance Use Disorder has been showing a rising trend all over the world including India. The project tested whether a Integrated community wide effort of Prevention and Awareness Groups (PAG) to manage substance use would have a greater effect on treatment attendance and drug abstinence than a de-addiction program alone.

ELIGIBILITY:
Inclusion Criteria:

* suburban, rural Population
* Drug and/or alcohol dependency (DSM-IV substance use disorders criteria)

Exclusion Criteria:

* Did not consent to participate
* Planning to move or relocate
* Severe mental disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2014-08; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Treatment attendance | Change from baseline to six month

SECONDARY OUTCOMES:
Drug abstinence | Change from baseline to six month

OTHER OUTCOMES:
Quality of Life assessed by General Health Questionnaire (GHQ) | Change from baseline to six months

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Murray, MA, Study Director — Goldington Family Centre; Neha Sharma, PhD, Principal Investigator — NMP Medical Research Institute; Amit Punia, LLB, Study Chair — NMP Medical Research Institute
Locations (1):
- GyanSanjeevani, Bai, Nawalgarh, Rajasthan, India